CLINICAL TRIAL: NCT06637982
Title: Extended Platelet Rich Fibrin in Mandibular Alveolar Ridge Splitting With Simultaneous Implant Placement
Brief Title: Extended Platelet Rich Fibrin in Mandibular Alveolar Ridge Splitting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0302024OS
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Ridge Splitting

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ridge splitting with allograft and pericardium membrane (Experimental)
  Interventions: Procedure: ridge splitting with the use of allograft and pericardium membrane
- ridge splitting with extended platelet rich fibrin (Experimental)
  Interventions: Procedure: ridge splitting with the use of extended platelet rich fibrin

INTERVENTIONS:
Procedure: ridge splitting with the use of allograft and pericardium membrane — ridge splitting with the use of allograft and pericardium membrane
  Arms: ridge splitting with allograft and pericardium membrane
Procedure: ridge splitting with the use of extended platelet rich fibrin — ridge splitting with the use of extended platelet rich fibrin
  Arms: ridge splitting with extended platelet rich fibrin

SUMMARY:
Thirty two healthy implants will be selected from the outpatient clinic of the oral and maxillofacial department of Mansoura university to be included in this study for replacement of lost posterior teeth with limited bone width.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years old and older.
* Patient's cooperation, motivation and good oral hygiene.
* Atrophic posterior mandible of horizontal alveolar dimension range between 3 - 6 mm at the crest, with minimum 10 mm vertical height from the alveolar crest to the superior border of the inferior alveolar canal.
* Absence of undercuts in buccal aspect of the ridge.
* Favorable occlusion and no parafunctional habits.
* Patients able to comply with the required recall visits.
* No gender preface in selection of the patients.
* Acceptable inter-arch space for the future prosthesis.

Exclusion Criteria:

* Any pathological condition at the site of surgery.
* Patients with systemic diseases that contra-indicate the surgical procedure such as uncontrolled diabetes mellitus, bleeding disorders, serious osseous disorders, and mental disorders.
* Patient taking drugs that could affect bone healing process as immunosuppressive drugs and bisphosphonates.
* Heavy smoking and alcoholism.
* Parafunctional habits such as bruxism and clenching.
* Signs of acute infection or pus discharge.
* Untreated periodontal disease or bad oral hygiene.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
implant stability | 9 months
  the stability of the implants will be evaluated by RFA with the Osstell Mentor device
alveolar ridge width | 9 months
  alveolar ridge width will be measured preoperative, immediate postoperative and after 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Mansoura, Egypt, Egypt